CLINICAL TRIAL: NCT01283555
Title: Comparative Safety Study of Pre-Filled Plastic and User-Filled Paper Vaginal Applicators With Candidate Microbicide, Tenofovir
Brief Title: Comparative Safety Study of Two Vaginal Applicators With Tenofovir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: CONRAD (Other); Profamilia, Santo Domingo, DR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PATH HS-522
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Results first posted 2012-06-22 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-06

CONDITIONS: Microbicide Applicator
Keywords: Microbicide, Applicator, Safety
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- User-Filled Applicator (Experimental)
  Interventions: Drug: Tenofovir
- Prefilled applicator (Other)
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir — Delivered using prefilled and user-filled applicator
  Other Names: TFV

SUMMARY:
The primary objective of this study is to compare the effect of two vaginal applicators, delivering the candidate microbicide Tenofovir, on symptoms and signs of irritation of the external genitalia, cervix and vagina as seen on colposcopy after seven days of twice daily use.

The secondary objectives are to:

1. Evaluate and compare the dosing accuracy and precision of the user-filled applicator and pre-filled applicator with the candidate microbicide, Tenofovir.
2. Compare the acceptability of the user-filled applicator with the pre-filled applicator.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 to 50, inclusive
* Pre-menopausal
* In good health as reported by individual
* Have regular menstrual cycles (24 to 35 days)
* Low risk for sexually transmitted infections (only one sexual partner in the last three months)
* Not pregnant or at risk of pregnancy (must either have had a tubal ligation, or currently be using a hormonal method of contraception)
* Negative on a urine pregnancy test
* Willing to abstain from sexual intercourse and masturbation during two 7-day periods when applicators are being used
* Willing to abstain from use of vaginal products during course of study (including douching, use of vaginal applicators for medication, lubrication, sex toys, other)
* Willing to follow procedural requirements of study
* Willing and able to provide informed consent for study participation
* Willing to provide investigator with phone number or address where she can be reached during the study

Exclusion Criteria:

* History of hysterectomy
* Pregnancy or within two months of last pregnancy outcome (delivery, spontaneous or induced abortion, medical or surgical management of ectopic pregnancy)
* Post-menopausal
* Breastfeeding
* Use of an intra-uterine device (IUD), cervical caps or diaphragm for contraceptive purposes
* Diagnosis or treatment for a sexually transmitted disease within the past 30 days;
* More than one sexual partner in the last 3 months
* Has had surgery on the external genitalia, vagina, or cervix within the past 3 months;
* Current or past use of any anti-retroviral therapies including but not limited to systemic Tenofovir (Viread®)
* Current or anticipated use of drugs on a daily basis that may reduce renal function (e.g. acyclovir or ibuprofen) or liver function (e.g. Tylenol)
* HIV positive at time of screening
* Hepatitis B surface antigen (HBsAg) positive at time of screening
* Positive test results for Neisseria gonorrhea, Chlamydia trachomatis, or Trichomonas vaginalis at time of screening.
* At baseline colposcopic exam (Visit 2), findings involving disruption of epithelium with disruption of blood vessels or deep disruption of epithelium alone. Any area of epithelium with bleeding will be considered deeply disrupted.
* Any abnormal finding on colposcopic exams which in the opinion of the investigator, precludes participation in the study
* At baseline exams, clinical symptoms or signs of vaginitis or vulvitis confirmed by a wet mount exam of the discharge. Note: If vaginitis or vulvitis is present at either baseline exam (visits 2 or 10), volunteer will be treated and rescheduled for new baseline exam one week after application of last treatment dose. If signs or symptoms are still present at the rescheduled baseline exam for Visit 2, the volunteer will not be enrolled into study. If signs or symptoms are still present at the rescheduled baseline exam for Visit 10, the volunteer will be discontinued from the study.
* Serum chemistry (glucose, creatinine, bilirubin, AST [aspartate aminotransferase] and ALT [alanine transaminase]) not within normal expected levels according to the specifications of the local laboratory.
* Hemoglobin, hematocrit and total white blood cell not within 15 % of lower and upper limit normal levels according to the specifications of the local laboratory.
* Participation in any other research study in the 30 days prior to screening and/or plans to participate in any other research study during the entire study duration.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Brache, Principal Investigator — Profamilia
Locations (1):
- Clinica Profamilia, Santo Domingo, Dominican Republic

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 26 January 2011 and ended on 10 March 2011. Recruitment was done at Clinica Profamilia, Santo Domingo, Dominican Republic. Healthy women, 18 to 50 years of age (inclusive), who attended the clinic for health care, who were not at risk for pregnancy, and at low risk of sexually transmitted infection were informed of the study.
Pre-assignment Details: 25 were enrolled in this study which used a cross-over design. Participants were randomized to order of applicator use.
Groups:
- User-Filled Applicator First, Then Prefilled: User-filled paper applicator (filled using a tube of Tenofovir 1% gel)used twice daily in first intervention period and prefilled applicator used twice daily in second intervention period (after washout period)
- Prefilled Applicator First, Then User-filled: Plastic applicator (prefilled with Tenofovir 1% gel) used twice daily in first intervention period and user-filled applicator used twice daily in second intervention period (after washout period)
Period: First Intervention
Arm/Group | User-Filled Applicator First, Then Prefilled | Prefilled Applicator First, Then User-filled
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: Washout Period of at Least 21 Days
Arm/Group | User-Filled Applicator First, Then Prefilled | Prefilled Applicator First, Then User-filled
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | User-Filled Applicator First, Then Prefilled | Prefilled Applicator First, Then User-filled
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to use the prefilled applicator first and the user-filled applicator first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  Dominican Republic | 25

OUTCOME MEASURES:

1. Secondary Outcome: Filled Volume
Description: At each dose delivery visit, the applicator was weighed, prior to vaginal insertion. For the user-filled applicator, the participant handed the applicator to the investigator after filling with gel from the multidose tube. The applicator was then weighed and returned to the participant for insertion. For the prefilled applicator, the participant inserted the plunger into the barrel, and then handed the applicator to the investigator for weighing.
Time Frame: 3 dose delivery measurements during 1 week of product use
Population: Per protocol all participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: ml
Units Other Than Participants: filled volume
Groups:
- User-Filled Applicator: paper applicator (filled using a tube of Tenofovir 1% gel)
- Prefilled Applicator: plastic applicator (prefilled with Tenofovir 1% gel)
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
Number analyzed (filled volume) | 75 | 75
ml | 4.22 (.24) | 4.11 (.07)

2. Secondary Outcome: Filling Precision (5% Range)
Description: A 5% range was calculated around the average filled volumes to determine how many applicators were filled within this range (+/-5% of average volume)
Time Frame: 3 dose delivery measurements during 1 week of product use
Population: Per protocol all participants were included in the analysis.
Measure: Number; unit: doses
Units Other Than Participants: volume of filled applicator
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
Number analyzed (volume of filled applicator) | 75 | 75
doses | 69 | 75

3. Secondary Outcome: Filling Precision (10% Range)
Description: A 10% range was calculated around the average filled volumes to determine how many applicators were filled within this range (+/-10% of average volume)
Time Frame: 3 dose delivery measurements during 1 week of product use
Population: Per protocol all participants were included in the analysis.
Measure: Number; unit: doses
Units Other Than Participants: volume of filled applicators
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
Number analyzed (volume of filled applicators) | 75 | 75
doses | 74 | 75

4. Secondary Outcome: Filling Accuracy (% of Target Dose)
Description: The target dose for Tenofovir gel in this study was 4.0ml, which is the volume of Tenofovir being used in current microbicide clinical trials. The filled volume for each applicator was compared with the intended target dose of 4.0ml.
Time Frame: 3 dose delivery measurements during 1 week of product use
Population: Per protocol all participants were included in the analysis.
Measure: Number; unit: % of target dose filled into applicator
Units Other Than Participants: volume of filled applicator
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
Number analyzed (volume of filled applicator) | 75 | 75
% of target dose filled into applicator | 105.5 | 102.8

5. Secondary Outcome: Dosing Volume (Expressed Volume)
Description: At each dose delivery visit, the applicator was weighed prior to vaginal insertion and after use. The volume of gel expressed was measured using the following data: weight of filled applicator, weight of emptied applicator, the average weight of an empty applicator, and gel density.
Time Frame: 3 dose delivery measurements during 1 week of product use
Population: Per protocol, all participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: ml
Units Other Than Participants: dosing volume
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
Number analyzed (dosing volume) | 75 | 75
ml | 3.83 (.35) | NA (NA) — As a result of an error in the interpretation of the user instructions, the dose delivery data for the prefilled applicator was not valid.

6. Secondary Outcome: Dosing Precision, 5% (Expressed Volume)
Description: A 5% range was calculated around the average expressed volume of 3.83ml to determine how many applicators delivered a dose within this range (+/-5% of average volume)
Time Frame: 3 dose delivery measurements during 1 week of product use
Population: Per protocol all participants were included in the analysis.
Measure: Number; unit: doses
Units Other Than Participants: dosing volume
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
Number analyzed (dosing volume) | 75 | 75
doses | 48 | NA — As a result of an error in the interpretation of the user instructions, the dose delivery data for the prefilled applicator was not valid.

7. Secondary Outcome: Dosing Precision, 10% (Expressed Volume)
Description: A 10% range was calculated around the average expressed volume of 3.83ml to determine how many applicators delivered a dose within this range (+/-10% of average volume)
Time Frame: 3 dose delivery measurements during 1 week of product use
Population: Per protocol all participants were included in the analysis.
Measure: Number; unit: doses
Units Other Than Participants: dosing volume
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
Number analyzed (dosing volume) | 75 | 75
doses | 64 | NA — As a result of an error in the interpretation of the user instructions, the dose delivery data for the prefilled applicator was not valid.

8. Secondary Outcome: Dosing Accuracy (% of Target Dose Delivered)
Description: The target dose for Tenofovir gel in this study was 4.0ml, which is the volume of Tenofovir being used in current microbicide clinical trials. The average dose delivered for each applicator was compared with the intended target dose of 4.0ml.
Time Frame: 3 dose delivery measurements during 1 week of product use
Population: Per protocol all participants were included in the analysis.
Measure: Number; unit: percent of target dose delivered
Units Other Than Participants: dosing volume
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
Number analyzed (dosing volume) | 75 | 75
percent of target dose delivered | 96 | NA — As a result of an error in the interpretation of the user instructions, the dose delivery data for the prefilled applicator was not valid.

9. Secondary Outcome: Number of Participants Reporting Applicator Easy to Fill
Description: Participants were asked to describe the process of filling the user-filled applicator.
  Response categories included "easy", "moderately difficult", and "difficult".
  Since "ease of filling" only applies to the user-filled applicator, this question was not applicable for the prefilled applicator.
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | User-Filled Applicator
Number analyzed (Participants) | 25
participants
  Easy | 25
  Moderately difficult | 0
  Difficult | 0

10. Secondary Outcome: Number of Respondents Reporting Confidence With Filling the User-filled Applicator
Description: Participants were asked when using the user-filled applicator, how confident did they feel that they at inserted the correct amount of gel into the applicator.
  Response categories included "very confident", "confident", and "not confident".
  (Note: this question does not apply to the prefilled applicator.)
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | User-Filled Applicator
Number analyzed (Participants) | 25
participants
  Very confident | 4
  Confident | 21
  Not confident | 0

11. Secondary Outcome: Reasons Given by Participants for Knowing When the Applicator Was Filled Correctly
Description: Participants were asked how did they know when the applicator was filled correctly (that is, with the right amount of gel). More than one answer was allowed.
  Response categories included "plunger automatically stopped", "the 'FULL' line was reached", and "other".
  Note: this question does not apply to the prefilled applicator.
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis. Each participant could identify multiple reasons. As a result, the number of units analyzed is greater than the number of participants.
Measure: Number; unit: participants
Units Other Than Participants: responses
Arm/Group | User-Filled Applicator
Number analyzed (Participants) | 25
Number analyzed (responses) | 29
participants
  Plunger automatically stopped | 9
  The fill line/arrow was reached | 18
  Other | 2

12. Secondary Outcome: Number of Participants Reporting Applicator Easy to Insert
Description: Participants were asked to describe the insertion of the applicator into the vagina for each applicator (user-filled and prefilled).
  Response categories included "easy", "moderately difficult", and "difficult".
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
participants
  Easy | 21 | 22
  Moderately difficult | 2 | 3
  Difficult | 2 | 0

13. Secondary Outcome: Number of Participants Reporting That the Gel Was Easy to Dispense
Description: Participants were asked to describe the dispensing of the gel into the vagina with each applicator (user-filled and prefilled).
  Response categories included "easy", "moderately difficult", and "difficult".
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
participants
  Easy | 24 | 23
  Moderately difficult | 1 | 2
  Difficult | 0 | 0

14. Secondary Outcome: Number of Participants Reporting Applicator Preference (User-filled or Prefilled) Across a Variety of Factors
Description: Participants were asked about their preference for either the user-filled or prefilled applicator with regard to several use factors as well as in relation to disposal, storage, and overall comfort and preference.
  Response categories included "user-filled", "prefilled", and "same".
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: responses
Groups:
- Same: no preference between user-filled or prefilled applicator
Arm/Group | User-Filled Applicator | Prefilled Applicator | Same
Number analyzed (Participants) | 25 | 25 | 25
responses
  Ease of use | 10 | 11 | 4
  Ease of insertion | 12 | 10 | 3
  Ease of dispensing gel | 8 | 8 | 9
  Ease of disposal | 19 | 0 | 6
  Ease of storage | 3 | 16 | 6
  Overall comfort | 11 | 10 | 4
  Overall applicator preference | 15 | 10 | 0

15. Secondary Outcome: Number of Participants Reporting That Applicator Was Comfortable to Use
Description: Participants were asked to describe the comfort of use for each applicator type(user-filled and prefilled).
  Response categories included "comfortable", "neutral", and "uncomfortable".
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
participants
  Comfortable | 19 | 20
  Neutral | 6 | 5
  Uncomfortable | 0 | 0

16. Secondary Outcome: Number of Participants Reporting Suggestions Regarding Ease of Use or Comfort
Description: Participants were asked if they could suggest ways that would make each applicator easier or more comfortable to use. Response categories were "yes" and "no". If yes, participants were asked to describe how they would make the applicator easier and/or more comfortable to use.
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
participants
  Yes | 7 | 5
  No | 18 | 20

17. Secondary Outcome: Number of Participants Reporting That the Instructions for Use Were Helpful
Description: For each applicator type, participants were asked if the instructions were helpful to you.
  Response categories were "yes" and "no".
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | User-Filled Applicator | Prefilled Applicator
Number analyzed (Participants) | 25 | 25
participants
  Yes | 25 | 25
  No | 0 | 0

18. Secondary Outcome: Number of Participants Reporting That Both Applicators Were Acceptable
Description: Participants were asked if both applicators were acceptable to them. Responses were either "yes" or "no".
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 25
participants
  Yes | 24
  No | 1

19. Secondary Outcome: Number of Participants Reporting That the Cost of the Applicator Would Influence Their Choice of Applicator
Description: Participants were asked if the cost of the applicator would influence their choice of applicator.
  Response categories were "yes", "no", and "maybe".
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 25
participants
  Yes | 6
  No | 12
  Maybe | 7

20. Primary Outcome: Number of Colposcopic Findings (Baseline and After One Week of Product Use)
Description: Comparison of colposcopic findings between baseline visits and after one week of twice-daily application of Tenofovir 1% gel with either a user-filled or prefilled applicator
Time Frame: 7 days
Population: The number of participants for analysis was determined by counting the number of participants with colposcopic findings and baseline and after one week of product use.
Measure: Number; unit: colposcopic findings
Units Other Than Participants: colposcopic findings
Groups:
- Baseline Colposcopic Findings: Number of colposcopic findings identified during baseline colposcopies for both study arms. Note: Since a participant can have more than one colposcopic finding, the number of colposcopic findings does not necessarily equal the number of participants with colposcopic findings.
- Colposcopic Findings After 7 Days of Product Use: Number of colposcopic findings identified during colposcopy after one week of twice daily product use (data from both study arms are combined). Note: Since a participant can have more than one colposcopic finding, the number of colposcopic findings does not necessarily equal the number of participants with colposcopic findings.
Arm/Group | Baseline Colposcopic Findings | Colposcopic Findings After 7 Days of Product Use
Number analyzed (Participants) | 25 | 25
Number analyzed (colposcopic findings) | 8 | 4
colposcopic findings
  Petechiae | 3 | 0
  Laceration external genitalia | 2 | 0
  Peeling cervic or vagina | 1 | 3
  Petechiae (iatrogenic) | 1 | 1
  Ecchymosis left lateral vaginal wall (iatrogenic) | 1 | 0
Statistical Analysis 1: Comparison: Baseline Colposcopic Findings vs Colposcopic Findings After 7 Days of Product Use; Fishers exact test was used to compare the frequency of non-iatrogenic colposcopic findings at baseline and follow-up visits (after one week of twice-daily product use); Test type: Superiority or Other; p = 0.4870, Fisher Exact — The p-value presented here represents a comparison of the total number of non-iatrogenic findings at baseline and after one week of product use

21. Secondary Outcome: Number of Participants Reporting That They Would Use the User-filled Applicator in the Future if it Came With a Gel for HIV Prevention
Description: Participants were asked if they would use the user-filled applicator in the future if it came with a gel that helped prevent HIV infection.
  Response categories included "yes", "no", and "in some circumstances".
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 25
participants
  Yes | 24
  No | 0
  In some circumstances | 1

22. Secondary Outcome: Number of Participants Reporting That They Would Not Want to Use the User-filled Applicator in the Future if it Came With a Gel for HIV Prevention
Description: Participants were asked if there were any reasons that they would not want to use this user-filled applicator in the future if it came with a gel that helped prevent HIV infection.
  Response categories included "yes", "no", and "in some circumstances".
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 25
participants
  Yes | 2
  No | 23
  In some circumstances | 0

23. Secondary Outcome: Number of Participants Reporting That They Would Recommend the User-filled Applicator for HIV Prevention
Description: Participants were asked if they would recommend the user-filled applicator to other women if it came with a gel that helped prevent HIV infection.
  Response categories included "yes", "no", and "in some circumstances".
Time Frame: Final study visit (after completing both study arms)
Population: All participants were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 25
participants
  Yes | 25
  No | 0
  In some circumstances | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were collected for the entire study period: January 26, 2011, to June 10, 2011.
Arm/Group | User-Filled Applicator | Prefilled Applicator
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 10/25 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | User-Filled Applicator (N=25) | Prefilled Applicator (N=25)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Common cold (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (2)
Tooth pain (Gastrointestinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to an error in the interpretation of the user instructions and resulting depth of plunger insertion into the barrel by the participants, the dose delivery data for the prefilled applicator were not valid.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators have agreed to provide drug sponsor with a copy of any draft manuscript or abstract for its review and comment at least thirty days prior to submission for publication and provide a copy of any draft presentation at least seven days in advance of any scientific meeting or conference.